CLINICAL TRIAL: NCT04538235
Title: Analgesic Non Inferiority of the Thoracic Bi-block Combining an Erector Spinae Muscle Plane Block and a Serratus Anterior Muscle Plane Block in Comparison With Thoracic Epidural for Video-Assisted Thoracic Surgery.
Brief Title: Analgesic Non Inferiority of the Thoracic Bi-block in Comparison With Thoracic Epidural for VATS.
Acronym: ANESSTEVATS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0473
Record Dates: First submitted 2020-09-02; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Erector Spinae Muscle Plane Block; Serratus Anterior Muscle Plane Block; Video-Assisted Thoracic Surgery; Lung Cancer; Pleural Diseases; Thoracic Epidural; Analgesia; Enhanced Recovery After Surgery
Keywords: regional anesthesia; video-assisted thoracic surgery
MeSH Terms: conditions — Lung Neoplasms; Pleural Diseases; Agnosia | interventions — Tea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bi-block (Serratus and erector spinae block) group: The Bi-block consisted in performing an ESP block followed by a SAP block on the side ipsilateral to the thoracic surgery. For the ESP block, 40 ml of Ropivacaine 2mg/ml were injected under the erector spinae muscle plane, at the level of the 4th thoracic vertebra. For the SAP block, 40 ml of Ropivacaine 2 mg/ml were injected under the serratus anterior muscle plane. The cumulative dose of Ropivacaine did not exceed 3 mg/kg.
  Regional anesthesia was performed before surgery.
  Interventions: Procedure: Thoracic Regional Analgesia
- Thoracic Epidural Analgesia (TEA) group: The thoracic epidural was performed according to a standardized protocol, with a Tuohy needle via the median puncture technique, at the level of T4-T5 intervertebral space. After a test dose of 2 to 3 ml of Lidocaine, 5 to 10 ml of a mixture of Ropivacaine 2 mg/ml and Sufentanil 0.5 µg / mL were injected. Epidural continuous administration was performed with the same mixture of anesthetic connected to a CADD Solis ™ pump set according to a PCEA protocol adapted to the patient's weight (continuous flow rate from 3 to 6 ml/h, self-administered bolus dose from 3 to 5 ml, refractory period 30 min).
  Regional anesthesia was performed before surgery.
  Interventions: Procedure: Thoracic Regional Analgesia

INTERVENTIONS:
Procedure: Thoracic Regional Analgesia — In the TEA group, a thoracic epidural was performed before VATS. In the Bi-block group, a SAP block associated with an ESP block were performed before surgical incision under general anesthesia.
  Other Names: Thoracic Epidural Analgesia; Bi-block, a regional anesthesia technique combining a serratus anterior block with an erector spinae block

SUMMARY:
Video-Assisted thoracic surgery (VATS) is the standard treatment for localized lung cancer. However, there is no consensus on analgesic management in patients undergoing VATS.

The aim of the study is to compare the analgesic efficacy of thoracic epidural with that a "Bi-block" combining an Erector Spinae muscle plane Block (ESP) and a Serratus Anterior Block (SAP) in patients undergoing VATS for lung or pleural surgery.

Our main hypothesis is that the analgesic efficacy of the Bi-block, assessed by morphine consumption, is not inferior to that provided by a thoracic epidural during the first 48 hours after VATS. We conducted a age, gender and type of surgery-matched retrospective cohort study in the Department of Thoracic Anesthesia of the Montpellier University Hospital (France).

ELIGIBILITY:
Inclusion Criteria:

* To be over 18.
* To be scheduled for VATS in the center of the study during the study period.
* Thoracic Epidural analgesia of Bi-block analgesia.

Exclusion Criteria:

* Chronic pain or opioid use before surgery (6 months).
* Postoperative hospitalization in ICU during the first two days.
* Postoperative surgical complication needing surgical revision during the first two days.
* Preoperative dementia or other psychiatric disease incompatible with VAS pain scoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each patient enrolled in the Bi-block group were matched by age, gender and type of surgery with two controls in the TEA group. Patients not-matched were secondarily excluded.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
cumulative morphine consumption on postoperative day 2 | postoperative day 2
  cumulative morphine consumption on postoperative day 2, including the morphine administered in Post anesthesia care unit (PACU), on postoperative day 0, 1 and 2.

SECONDARY OUTCOMES:
non-opioid analgesics consumption on postoperative day 2 | postoperative day 2
  Paracetamol, Tramadol, Ketoprofen, Nefopam cumulative consumption on POD 2.
Pain assessed by visual analog pain scale (VAS) | up to postoperative day 2
  mean VAS, maximal VAS, number of events with a VAS > 3
Urinary retention | up to postoperative day 2
hypotension | up to postoperative day 2
pleural drain duration | up to postoperative day 2
duration of hospitalization | up to postoperative day 2
occurrence of prurit | up to postoperative day 2

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Sentenac, MD, Principal Investigator — Montpellier University Hospital; Pascal H Colson, MD, PhD, Study Chair — Montpellier University Hospital
Locations (1):
- Intensive Care Unit, D - University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided